CLINICAL TRIAL: NCT00034619
Title: A Phase 2 Trial of ALIMTA (LY231514, Pemetrexed) Plus Oxaliplatin Administered Every 21 Days for First-Line Treatment of Patients With Advanced Colorectal Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Purpose: Treatment
Other Study IDs: 5142; H3E-MC-JMEP
Record Dates: First submitted 2002-05-01; First posted 2002-05-02 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Pemetrexed; Oxaliplatin

INTERVENTIONS:
Drug: ALIMTA
Drug: Oxaliplatin

SUMMARY:
The purpose of this study is to assess the antitumor activity of ALIMTA plus Oxaliplatin combination therapy in patients with previously untreated advanced colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary cancer of the colon or rectum
* Must have measurable disease
* Must be able to comply with study procedure

Exclusion Criteria:

* Prior chemotherapy for advanced disease
* Pregnancy or lactation
* Candidates for surgical resection of one or more metastatic foci
* Second primary cancer
* Inability to take folic acid or vitamin B12

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - "For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559)", Huntsville, Alabama
  - "For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559)", Pittsfield, Massachusetts
  - "For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559)", Kalamazoo, Michigan
  - "For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559)", Latham, New York
  - "For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559)", Asheville, North Carolina
  - "For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559)", Goldsboro, North Carolina
  - "For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559)", Hendersonville, North Carolina
  - "For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559)", Winston-Salem, North Carolina
  - "For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559)", Columbus, Ohio
  - "For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559)", Bend, Oregon
  - "For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559)", Portland, Oregon
  - "For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559)", Philadelphia, Pennsylvania
  - "For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559)", Pittsburgh, Pennsylvania
  - "For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559)", Reading, Pennsylvania
  - "For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559)", Charleston, South Carolina
  - "For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559)", Ivins, Utah
  - "For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559)", Ogden, Utah
  - "For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559)", Provo, Utah
  - "For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559)", St. George, Utah
  - "For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559)", Bellevue, Washington
  - "For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559)", Seattle, Washington
  - "For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559)", Spokane, Washington